CLINICAL TRIAL: NCT06113536
Title: Evaluation of Meniscal Extrusion by Dynamic Ultrasonography in Patients With Ostearthritis and Comparison With Magnetic Resonance Imaging Study.
Brief Title: Evaluation of Meniscal Extrusion by Dynamic Ultrasonography in Patients With Ostearthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-MEN
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Meniscus Disorder
Keywords: dynamic ultrasonography; Nuclear magnetic resonance imaging; Meniscal extrusion; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is a diagnostic, open-label, single-center interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasonographic evaluation (Experimental): Ultrasonographic evaluation for assessment of possible meniscal extrusion
  Interventions: Diagnostic Test: Ultrasonographic evaluation

INTERVENTIONS:
Diagnostic Test: Ultrasonographic evaluation — Ultrasonographic evaluation for assessment of possible meniscal extrusion

SUMMARY:
This is a diagnostic, open-label, single-center interventional study. The aim of the study is to evaluate the relationship between medial and lateral meniscus extrusion determined by dynamic ultrasound study and bone edema assessed by MRI study in patients with knee OA.

As a secondary objective, the correlation of the above parameters with the patient's symptomatology assessed by subject clinical questionnaires will be evaluated.

DETAILED DESCRIPTION:
Patients with a diagnosis of knee OA will be included in a study involving evaluation of the correlation between meniscal extrusion assessed by dynamic ultrasonography and bone edema assessed on MRI. A total of 202 patients will be included, who, after providing their signed informed consent to participate in the study, will undergo dynamic ultrasonography. After giving signed consent to participate in the study, the patient will undergo the following examinations::

* ultrasound evaluation for assessment of possible meniscal extrusion;
* At the same time as the ultrasound examination, subjective questionnaires will be administered to patients.Recent radiological examinations of the patients or from the patient's medical record will be collected during or before the diagnostic investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. Signs and symptoms of degenerative pathology of knee cartilage;
3. Patients with Radiographic (X-ray or MRI) signs of OA (K-L grade 0-4); 3.
4. Cooperative patients with pain that does not prevent orthostatism
5. Ability and consent of patients to actively participate in clinical follow-up;
6. Recently performed MRI (maximum 1 month).

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients undergoing intra-articular infiltration of other substance in the previous 6 months;
3. Patients undergoing knee surgery in the previous 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with a history of total/subtotal meniscectomy;
7. Patients with symptomatology such that a dynamic examination in orthostatism is not possible; 7.
8. Patients abusing alcoholic beverages, drugs or medications;
9. Body Mass Index > 40;
10. Pregnant or lactating women;
11. Patients with axis deviation > 5°.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Meniscal extrusion | baseline
  Meniscal extrusion in clinostatism and orthostatism, assessed in millimeters (mm) or percent meniscal extrusion relative to tibial margin, and difference between the two measurements

SECONDARY OUTCOMES:
IKDC-Subjective Score (Subjective International Knee Documentation Committee) | baseline
  The IKDC-Subjective Score (Subjective International Knee Documentation Committee) is a subjective, knee-specific rating scale.The questionnaire examines 3 categories: symptoms, sports activity, and knee function. The response "Unable to perform any of the above activities due to knee pain" receives a score of 0 while the response "Very strenuous activities like jumping or pivoting as in basketball or soccer" receives a score of 4. This is how item 1, which is related to the highest level of activity without significant pain, is scored. For item 2, which asks about the frequency of pain in the last four weeks, the responses "Constant" and "Never" receive scores of 0 and 10, respectively
KOOS Score ( Knee Injury and Osteoarthritis Outcome score) | baseline
  The full questionnaire consists of five subscales and they cover: pain (9 items), symptoms (7 items of which two relate to stiffness), functions and activities of daily living (17 items) physical function, sports activities and leisure (5 items) and quality of life in relation to the knee (4 items). All items in the relevant subscales have the same response mode, use a 5-point Likert scale, and each question is assigned a score from 0 to 4, where 0 indicates "no difficulty" and 4 "a severe difficulty). Score range 0-100 for each subscale
VAS-dolore (Visual Analogue Scale) | baseline
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable."
Tegner Activity Level Scale | baseline
  The Tegner Activity Level Scale: allows the estimation of a subject's motor activity level with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as soccer at the national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders.
EQ-VAS | baseline
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable."
Objective parameters - Circumferences | baseline
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis.The measurement will be taken by the orthopedist by meter and will be reported in centimeters
Objective parameters- Range of Motion | baseline
  Evaluation of the Range of Motion for comparative analysis. Range of motion (ROM) is a term used to describe how far you can move a joint or muscle in various directions. It is used to measure how much you can move a joint on your own (active ROM) or with the assistance of someone else (passive ROM).Range of motion is measured using a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Andriolo, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Englund M, Guermazi A, Roemer FW, Aliabadi P, Yang M, Lewis CE, Torner J, Nevitt MC, Sack B, Felson DT. Meniscal tear in knees without surgery and the development of radiographic osteoarthritis among middle-aged and elderly persons: The Multicenter Osteoarthritis Study. Arthritis Rheum. 2009 Mar;60(3):831-9. doi: 10.1002/art.24383. PMID 19248082
- [Background] Podlipska J, Guermazi A, Lehenkari P, Niinimaki J, Roemer FW, Arokoski JP, Kaukinen P, Liukkonen E, Lammentausta E, Nieminen MT, Tervonen O, Koski JM, Saarakkala S. Comparison of Diagnostic Performance of Semi-Quantitative Knee Ultrasound and Knee Radiography with MRI: Oulu Knee Osteoarthritis Study. Sci Rep. 2016 Mar 1;6:22365. doi: 10.1038/srep22365. PMID 26926836
- [Background] Ozdemir M, Turan A. Correlation Between Medial Meniscal Extrusion Determined by Dynamic Ultrasound and Magnetic Resonance Imaging Findings of Medial-Type Knee Osteoarthritis in Patients With Knee Pain. J Ultrasound Med. 2019 Oct;38(10):2709-2719. doi: 10.1002/jum.14976. Epub 2019 Mar 4. PMID 30828848
- [Background] Felson DT, McLaughlin S, Goggins J, LaValley MP, Gale ME, Totterman S, Li W, Hill C, Gale D. Bone marrow edema and its relation to progression of knee osteoarthritis. Ann Intern Med. 2003 Sep 2;139(5 Pt 1):330-6. doi: 10.7326/0003-4819-139-5_part_1-200309020-00008. PMID 12965941
- [Background] Wang Y, Wluka AE, Pelletier JP, Martel-Pelletier J, Abram F, Ding C, Cicuttini FM. Meniscal extrusion predicts increases in subchondral bone marrow lesions and bone cysts and expansion of subchondral bone in osteoarthritic knees. Rheumatology (Oxford). 2010 May;49(5):997-1004. doi: 10.1093/rheumatology/keq034. Epub 2010 Feb 24. PMID 20181669